CLINICAL TRIAL: NCT02004743
Title: Program Development in Guideline Development, Early Recognition and Specialized Treatment of Post Traumatic Stress Disorder (PTSD) at Sunnybrook Health Sciences Center, Canada's Largest Trauma Center
Brief Title: Early Prevention of Post Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 258-2012
Record Dates: First submitted 2013-02-22; First posted 2013-12-09 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Early Intervention; Prevention; Risk Factors; Exposure Therapy; Psychoeducation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Methods; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Other): Treatment as Usual
  Interventions: Other: Treatment as usual
- Intervention (Other): Psychological management guidelines + patient education
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Psychological guidelines and PET
  Patients will receive questionnaires at recruitment, 1 month, 3 months and 6 months based on the timeline of Diagnostic and Statistical Manual (DSM) -IV criteria for PTSD.
  Arms: Intervention
Other: Treatment as usual — Participants will experience treatment as usual.
  Patients will receive questionnaires at recruitment, 1 month, 3 months and 6 months based on the timeline of Diagnostic and Statistical Manual (DSM) -IV criteria for PTSD
  Arms: Control

SUMMARY:
Sunnybrook Health Sciences Centre is Canada's largest trauma centre, treating 1,100 patients annually. A traumatic experience can lead to post-traumatic stress disorder, which increases hospital stays, emergency visits and disability. Despite developing leadership to manage a "Code Orange" mass trauma, Sunnybrook lacks guidelines in the psychological management of patients who have experienced trauma. The department of psychiatry currently holds a Traumatic Brain Injury clinic and PTSD services for youth but lacks both immediate intervention, prevention and adult services. This research will enable us to gain best evidence expertise to develop guidelines as well as a sustainable PTSD treatment program, with clear outcomes to assess effectiveness, psychiatric morbidity, use of healthcare, disability and substance abuse.

The five world-expert-consensus intervention resilience based principles will be operationalized in guidelines for the management of trauma patients, their caregivers and in routine nursing and trauma team care from the Emergency to the ward, and discharge, through to outpatient care. It is hypothesized that this will improve the psychological recovery of patients at risk of developing PTSD after a traumatic injury. In addition, early screening and intervention for increased risk of PTSD will be implemented one month after the trauma. It is hypothesized that such trauma informed psychological management, early screening and expert treatment using prolonged exposure will reduce hospital stays, functional disability, as well as longer-term psychiatric morbidity, including substance abuse.

DETAILED DESCRIPTION:
The study is a longitudinal interventional study, with a control group who have treatment for their trauma with no guidelines for psychological management, staff training, patient and family intervention/education. In the intervention group, who will have all of the above, participants will be stratified according to risk factors for PTSD and randomized 1:1 in "low risk" and "at risk" groups-those who will have a prolonged exposure intervention and those who will not.

ELIGIBILITY:
Inclusion Criteria:

* undergone severe physical trauma within the last 3 days
* An abbreviated Injury Severity score of 1-3

Exclusion Criteria:

* 14 years of age or younger
* an inability to communicate sufficiently in English
* A diagnosis of psychosis, mental retardation and/or autism

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Presence & severity of PTSD symptoms | 1 month, 3 months & 6 months
  The aim of the study is to observe whether there's a presence and severity (if applicable) of Posttraumatic symptoms in patients who've received the intervention, compared to those who have not.
  Presence and severity of PTSD symptoms will be measured by:
  * follow-up at 1 month, 3 months & 6 months which involve specific PTSD self-report symptom measures: PTSD Symptom Scale
  * Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorder (SCID) Semi-structured interview performed at 6 months either over the phone or in person
Depressive symptoms | recruitment, 1 month, 3 months & 6 months
  The Beck Depression Inventory - Second Edition (BDI-II) will be used at recruitment, 1 month, 3 months, and 6 months follow-up to measure the presence and/or change in depressive symptoms of the patient.

SECONDARY OUTCOMES:
Anxiety & dissociation symptoms | recruitment & 1 month
  Patients will be assessed for anxiety and dissociation symptoms at recruitment and follow-up at 1 month with the Stanford Acute Stress Reaction Questionnaire (SASRQ).
Change in patient health & well-being | 6 months
  The Short Form (36) Health Survey (SF-36v2) will be used at 6 months follow-up to assess a patient's health and/or disability.
Change in substance use | recruitment, 1 month, 3 months & 6 months
  PTSD is highly correlated with substance use. By implementing a preventative intervention, one aim is to reduce overall substance use. This will be assessed using the Alcohol Use Disorders Identification Test (AUDIT) and the Drug Abuse Screening Test (DAST) at recruitment, 1 month, 3 months and 6 months.
Presence & severity of trauma related thoughts and beliefs | 1 month, 3 months & 6 months
  follow-up at 1 month, 3 months & 6 months which involve specific PTSD self-report symptom measures: The Posttraumatic Cogntions Inventory (PTCI)
Self-esteem | recruitment, 1 month, 3 months & 6 months
  The Rosenberg Self-Esteem Scale (RSES) will be used at recruitment, 1 month, 3 months, and 6 months follow-up to measure any change in the patient's self-esteem over time.
Locus of Control | recruitment, 1 month, 3 months & 6 months
  The Internal Control Index (ICI) will be used at recruitment, 1 month, 3 months, and 6 months follow-up to measure any changes with a patient's Locus of Control, the extent to which they feel they can control the events that occur to them.
Self-efficacy | recruitment, 1 month, 3 months & 6 months
  The Self-Efficacy Scale will be used at recruitment, 1 month, 3 months & 6 months follow-up to asses any changes in a patient's self-efficacy/personal competence.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Ellis, Dr., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided